CLINICAL TRIAL: NCT04952194
Title: Clinical Study of Stalevo in the Treatment of Early Parkinson's Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0279
Record Dates: First submitted 2021-06-03; First posted 2021-07-07 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Stalevo; entacapone; Levodopa; Carbidopa

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stalevo group (Experimental): Stalevo is taken five times a day, three hours apart. Compare the incidence of dyskinesia.
  Interventions: Drug: Stalevo
- Control group (Active Comparator): Carbidopa and Levodopa Sustained-release Tablets is taken five times a day, three hours apart. Compare the incidence of dyskinesia.
  Interventions: Drug: Carbidopa and Levodopa Controlled Release Tablets

INTERVENTIONS:
Drug: Stalevo — The dose of Stalevo initially ranges from (Levodopa/Carbidopa/Entacapone) 50/12.5/200 mg 3 times a day to a target dose of 100/25/200 mg 5 times a day, with an interval of 3 hours. No other anti-Parkinson's disease drugs are added.
  Other Names: Entacapone, Levodopa and Carbidopa Tablets
  Arms: Stalevo group
Drug: Carbidopa and Levodopa Controlled Release Tablets — The dose of Carbidopa and Levodopa Controlled Release Tablets initially ranges from (Levodopa/Carbidopa) 50/12.5mg 3 times a day to a target dose of 100/25 mg 5 times a day, with an interval of 3 hours. No other anti-Parkinson's disease drugs are added.
  Arms: Control group

SUMMARY:
The main goal of PD research is to develop disease-modifying drugs to delay or prevent the underlying neurodegenerative process. Levodopa, as the gold standard for PD treatment, is associated with the occurrence of motor complications. Many previous studies have confirmed that Stalevo can reduce the side effects of levodopa alone. Moreover, the effects of Stalevo on the treatment of PD patients have been extensively studied, but the efficacy of Stalevo in early PD patients has been less studied. Therefore, it is necessary to further study the treatment of early PD with Stalevo, and observe whether increasing the number of medication can reduce the occurrence of dyskinesis. The research results will help to deepen the understanding of Stalevo in the treatment of early PD and its clinical efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the trial and sign the informed consent
* The enrolled patients were 30 to 70 years old, diagnosed as primary Parkinson's disease according to the 2015 MDS Parkinson's disease diagnostic criteria, H-Y grade <3, and the onset time was less than 5 years
* Patients can take stable dopamine receptor agonists or other anti-Parkinson's disease drugs (drugs have not been adjusted in the past 4 weeks), and have not used amantadine or entacapone within 1 year.

Exclusion Criteria:

* Atypical Parkinsonism and Secondary parkinsonism

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The occurrence and frequency of dyskinesia of participants in two groups were assessed by blind method. | 1 year
  The duration of the study is 96 weeks. Follow-up: Baseline, 4 weeks, 8 weeks, 12 weeks, 24 weeks, 36 weeks, 48 weeks, 60 weeks, 72 weeks, 84 weeks, 96 weeks. At each visit, the doctor performs a blind assessment of dyskinesia. The proportion of patients with no dyskinesias in the two groups at each visit was recorded. The Kaplan-Meier line was used to analyze the relationship between the drug and the occurrence of dyskinesia.
The Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) of participants in two groups were assessed by blind method. | 1 year
  At each visit, the patient completed the MDS-UPDRS. The doctor performs a blind assessment of MDS-UPDRS parts II, III, and IV. MDS-UPDRS part II, Motor Experiences of Daily Living (13 items); part III, Motor Examination (33 items); and part IV, Motor Complications. (6 items). All items have five response options with uniform anchors of 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. The more severe the symptoms, the higher the score.
The 9-Item Wearing-Off Questionnaire （WOQ-9） score of participants in two groups were assessed by blind method. | 1 year
  During the double-blind period, subjects completed WOQ-9 at each visit. WOQ-9 was used to assess symptoms of wearing-off. The nine symptoms include tremor, anxiety, mood changes, slowness of movement, reduced dexterity, general stiffness, pain/aching, slowness of thinking , and muscle cramping. The presence of one of these symptoms and relief after the next dose is indicative of wearing-off.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affilliated Hospital Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No